CLINICAL TRIAL: NCT06915974
Title: Comparison Between Interleukin 6 and Procalcitonin in Detecting Sepsis and Incidence of Mortality in Burn ICU Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMASU MS 10/2024/2025
Record Dates: First submitted 2025-02-14; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Burns; Sepsis; Septic Shock; Death
MeSH Terms: conditions — Burns; Sepsis; Shock, Septic; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Burn ICU patients (Experimental): Interleukin 6 and procalcitonin will be sampled for all patients on days 1, 3, 7, and 10. Treatment plan will be initiated to all patients according to the burn ICU protocol.
  Interventions: Diagnostic Test: Interleukin 6

INTERVENTIONS:
Diagnostic Test: Interleukin 6 — Interleukin 6 and procalcitonin will be sampled for all patients on days 1, 3, 7, and 10
  Other Names: Procalcitonin

SUMMARY:
The investigators will compare the efficacy of Interleukin-6 (IL-6) as a better indicator than procalcitonin in burn patients with sepsis or septic shock regarding success of treatment and early ICU discharge.

DETAILED DESCRIPTION:
Interleukin 6 and procalcitonin will be sampled for all patients on days 1, 3, 7, and 10.

Treatment plan will be initiated to all patients according to the burn ICU protocol.

According to the lab results, interleukin 6 and procalcitonin will guide the investigators to take decisions regarding clinical improvement and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute burn admitted to burn ICU within 24 hours from the burn incidence.
* patients with burn percentage of 25% to 50% of total body surface area
* patients with second to third degree burns
* ASA 1 and ASA 2 patients

Exclusion Criteria:

* Burn percentage more than 50% or less than 25% of total body surface area
* Having autoimmune diseases
* Cancer patients
* ASA 3 and ASA 4 patients

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of sepsis and septic shock | From day 1 to day 10 in burn ICU
  Prediction of occurrence of sepsis and septic shock

SECONDARY OUTCOMES:
Length of ICU stay | One month after ICU admission
  Response to treatment and length of ICU stay for over one month

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Elsayed, M.B.B.CH, Principal Investigator — Anaesthesia, intensive care, and pain management resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once the study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2026
Access Criteria: Free